CLINICAL TRIAL: NCT06409949
Title: MitoQ Treatment of Claudication: Myofiber and Micro-vessel Pathology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0053-23-EP
Record Dates: First submitted 2024-04-17; First posted 2024-05-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Biopsy, Needle

STUDY DESIGN:
Intervention Model Description: Patients with peripheral artery disease and claudication will participate in a double-blind, randomized, placebo-controlled trial with two parallel arms. Patients will be randomized 2:1 to receive either a daily oral dose of 40 mg MitoQ or matched placebo for six months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, randomized, placebo-controlled trial with two parallel arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Active Comparator): Participants will be placed on a 24-week regimen of oral dosing with MitoQ. The patients will take two 20 mg caps of MitoQ on empty stomach, each morning
  Interventions: Diagnostic Test: Walking assessment; Other: QOL Survey; Diagnostic Test: Ankle pressure at rest and after stress; Diagnostic Test: Muscle Oxygen; Diagnostic Test: Serum MitoQ Level; Procedure: Needle Biopsy
- Placebo (Placebo Comparator): The patients will take two identical caps of matched placebo on empty stomach, each morning
  Interventions: Diagnostic Test: Walking assessment; Other: QOL Survey; Diagnostic Test: Ankle pressure at rest and after stress; Diagnostic Test: Muscle Oxygen; Diagnostic Test: Serum MitoQ Level; Procedure: Needle Biopsy

INTERVENTIONS:
Diagnostic Test: Walking assessment — Participating patients will undergo the following evaluations at baseline and after six months of treatment with MitoQ or placebo:
  Assessment of walking impairment: Evaluation of treadmill maximum walking distances, six-minute walking distance, and daily physical activity (average steps taken daily)
Other: QOL Survey — Assessment of quality of life: Survey of Quality of life with the Walking Impairment Questionnaire and Short Form 36
Diagnostic Test: Ankle pressure at rest and after stress — Assessment of leg hemodynamics: Evaluation of post-occlusive ankle pressure and ankle/brachial index
Diagnostic Test: Muscle Oxygen — Evaluation of calf muscle heme oxygen saturation
Diagnostic Test: Serum MitoQ Level — Evaluation of serum concentrations of MitoQ
Procedure: Needle Biopsy — Needle biopsy of the calf muscle

SUMMARY:
In our research, we are delving into whether taking MitoQ for six months can improve the symptoms and function of people diagnosed with peripheral artery disease, especially those who suffer from leg pain while walking, known as intermittent claudication. We will be checking if MitoQ helps people with claudication walk better, be more active every day, feel better about their lives, and if it enhances the health of their leg muscles.

DETAILED DESCRIPTION:
This study will investigate whether taking MitoQ for six months can improve the walking ability, daily activity levels, and quality of life of people with claudication (leg pain) caused by peripheral artery disease (PAD). We'll also look at how MitoQ affects their calf muscles.

Here's what we'll be checking:

Muscle health: We'll examine muscle tissue samples under a microscope to see if MitoQ improves muscle health and function.

Body chemistry: We'll check blood tests to see if MitoQ affects overall health markers.

Mitochondrial health: We'll see if MitoQ reduces damage to mitochondria (the cell's powerhouses) and helps the body get rid of damaged ones. We'll also see if it improves how well mitochondria function.

Blood flow: We'll measure blood flow in the legs and see if MitoQ improves the function of tiny blood vessels in the calf muscles.

In short, we want to see if MitoQ can improve various aspects of health in people with claudication and PAD, and if these improvements are linked to better functioning mitochondria in their muscles.

ELIGIBILITY:
Inclusion Criteria:

1. a positive history of chronic claudication
2. exercise-limiting claudication established by history and direct observation during a screening walking test administered by the evaluating vascular surgeon
3. documented lower extremity arterial occlusive disease based on ankle/brachial index measurements and/or arterial imaging
4. stable blood pressure, lipid and diabetes regimens and risk factor control for 6 weeks.

Exclusion Criteria:

1. rest pain or tissue loss due to PAD (Fontaine stage III and IV)
2. acute lower extremity ischemic event
3. walking capacity significantly and primarily limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Walking Impairment: maximum treadmill distance | Before and After 6 months of treatment with MitoQ or placebo
  Evaluation of maximum walking distance on treadmill until participant chooses to stop due to pain in his legs.

SECONDARY OUTCOMES:
Walking Impairment: 6 minute distance | Before and after 6 months of treatment with MitoQ or placebo
  Evaluation of maximum walking distance the participant can walk over 6 minutes in hallway.
Walking Impairment: initial claudication treadmill distance | Before and after 6 months of treatment with MitoQ or placebo
  Evaluation of walking distance on treadmill until participant starts experiencing claudication pain in his legs.
Walking Impairment: daily physical activity | Before and after 6 months of treatment with MitoQ or placebo
  Measurement of average steps taken daily using a pedometer
Walking Impairment Questionnaire | Before and after 6 months of treatment with MitoQ or placebo
  Walking Impairment Questionnaire: There are 14 questions across three categories of walking distance, walking speed and stair climbing.
  The WIQ is graded on a scale of 0-4; 0 represents no difficulty; 4 represents inability to walk. 0 score represents no difficulty, 1 score is slight difficulty, 2 score is some difficulty, 3 score is much difficulty, 4 score is unable to complete the task in question.
Walking Impairment Short Form-36 | Before and after 6 months of treatment with MitoQ or placebo
  Walking Impairment Short Form-36 - (The Short Form 36 Health Survey Questionnaire) has 8 scale (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health) that measures quality of life. The SF-36 scoring ranges from 0-100. Higher scores indicate better health; lower scores indicate more disability.
Leg hemodynamics ankle/brachial index at rest and after stress | Before and after 6 months of treatment with MitoQ or placebo
  Evaluation of ankle/brachial index at rest and after stress. The ankle-brachial index test compares the blood pressure measured at the ankle with the blood pressure measured at the arm. A care provider measures your blood pressure in both arms and both ankles. This is done using an inflatable cuff and a hand-held ultrasound device. The device uses sound waves to detect blood flow and allows the pulse in the ankle arteries to be heard after the cuff is deflated.
  The test will be done first with you resting and then under stress. The stress will be produced by a blood pressure cuff placed around the lower thigh and the cuff being inflated to block blood flow to your calf and foot for five minutes.The cuff is then deflated, allowing blood to flow back into the leg.
Leg hemodynamics muscle heme-oxygen (StO2) | Before and after 6 months of treatment with MitoQ or placebo
  Evaluation of the level of oxygen in your calf muscle at rest and during during exercise. StO2 is measured with a wireless, probe placed on the skin of your calf.
Calf muscle cell damage | Before and after 6 months of treatment with MitoQ or placebo
  In the small tissue sample (biopsy) from your calf muscle we will look at the damage of the muscle cells by oxidative stress and the way the shape and size of the cells changes. This will be measured with quantitative widefield fluorescence microscopy.
Calf muscle mitochondria function and damage | Before and after 6 months of treatment with MitoQ or placebo
  In the small tissue sample (biopsy) from your calf muscle we will look at the function and possible damage of the mitochondria in your muscle cells. Mitochondria are the powerhouses of your cells. We'll see if they're working properly or damaged.This will be measured with high-resolution respirometry, quantitative widefield fluorescence microscopy, 2-dimensional gel electrophoresis and mass spectrometry.
Calf muscle fibrosis | Before and after 6 months of treatment with MitoQ or placebo
  In the small tissue sample (biopsy) from your calf muscle we will look at the amount of scarring (fibrosis) and measure if there is there any scar tissue buildup in the muscle.This will be measured with high-resolution respirometry, quantitative widefield fluorescence microscopy and with multiSpectral wide-field microscopy.
Calf muscle inflammation | Before and after 6 months of treatment with MitoQ or placebo
  In the small tissue sample (biopsy) from your calf muscle we will measure the inflammation present in the muscle.This will be measured with quantitative widefield fluorescence microscopy and enzyme-linked immunosorbent assay.
Calf muscle blood vessel health | Before and after 6 months of treatment with MitoQ or placebo
  In the small tissue sample (biopsy) from your calf muscle we will check how well the tiny blood vessels inside your muscle are working and if they are damaged and how much.This will be measured with videomicroscopy of calf muscle micro-vessel vasomotor function, high-resolution respirometry and quantitative widefield fluorescence microscopy.
Level of MitoQ in the blood and the muscle | After 6 months of treatment with MitoQ or placebo
  In the blood sample and the muscle sample we will collect from you we will check the level of MitoQ. This will be measured with mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Iraklis Pipinos, MD, Principal Investigator — University of Nebraska
Locations (1):
- VA Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No